CLINICAL TRIAL: NCT01265446
Title: A Randomized, Double-blind, Parallel Group, Single-dose Study of the Efficacy of Lidocaine 8 mg + Cetylpyridinium Chloride (CPC) 2 mg Fixed Combination Lozenges on Sore Throat Pain Intensity Compared to Lozenges Containing Lidocaine 1 mg and CPC 2 mg in Subjects With Sore Throat Due to Upper Respiratory Tract Infection.
Brief Title: Efficacy and Safety of a Sore Throat Lozenge Containing Lidocaine and Cetylpyridinium Chloride in Patients With Sore Throat Due to a Common Cold.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 075-A-301; 2010-021653-39 (EudraCT Number)
Record Dates: First submitted 2010-12-20; First posted 2010-12-23 (Estimated); Results first posted 2012-07-26 (Estimated); Last update posted 2013-04-24 (Estimated); Status verified 2013-04

CONDITIONS: Sore Throat Due to a Common Cold
Keywords: Sore throat, upper respiratory tract infection, lozenge with lidocaine and cetylpyridinium chloride.
MeSH Terms: conditions — Pharyngitis; Respiratory Tract Infections | interventions — Lidocaine; cytidylyl-(3'-5')-cytidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lidocaine 8mg +CPC 2mg (Experimental): one single dose
  Interventions: Drug: Lidocaine 8mg + CPC 2mg
- Lidocaine 1mg + CPC 2mg (Active Comparator): one single dose
  Interventions: Drug: Lidocaine 1mg + CPC 2mg

INTERVENTIONS:
Drug: Lidocaine 8mg + CPC 2mg — one single dose
  Arms: Lidocaine 8mg +CPC 2mg
Drug: Lidocaine 1mg + CPC 2mg — one single dose
  Arms: Lidocaine 1mg + CPC 2mg

SUMMARY:
This study will compare the efficacy and safety of a single dose of a lidocaine 8 mg + cetylpyridimium chloride (CPC) 2 mg lozenge with a single dose of a lidocaine 1 mg + CPC 2 mg lozenge in the treatment of sore throat due to a common cold.

ELIGIBILITY:
Inclusion Criteria:

* Patients with sore throat due to an upper respiratory tract infection, with recent onset (within 48 hours)
* Sore throat of at least moderate pain intensity

Exclusion Criteria:

* - History of hypersensitivity to any of the study drugs and listed excipients or to drugs of similar chemical classes
* Evidence of mouth breathing or severe coughing
* Evidence of overt oropharyngeal bacterial or fungal infection or evidence of lower respirator tract infection
* Severe renal, liver or cardiac impairment
* Severe lung disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2010-12; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Investigator, Principal Investigator — SocraTec R&D GmbH
Locations (1):
- Socratec, Erfurt, Germany

REFERENCES:
- [Derived] Donath F, Mallefet P, Garreffa S, Furcha R. Efficacy of 8 mg lidocaine and 2 mg cetylpyridinium chloride (CPC) fixed-combination lozenges on sore throat pain intensity compared with 1 mg lidocaine and 2 mg CPC fixed-combination lozenges in subjects with sore throat due to upper respiratory tract infection: a randomized double-blind parallel-group single-dose study. Trials. 2018 Dec 12;19(1):679. doi: 10.1186/s13063-018-3077-6. PMID 30541606

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 14 Dec 2010 to 5 Apr 2011
Period: Overall Study
Arm/Group | Lidocaine 8mg +CPC 2mg | Lidocaine 1mg + CPC 2mg
Started | 125 | 125
Completed | 124 | 125
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lidocaine 8mg +CPC 2mg | Lidocaine 1mg + CPC 2mg | Total
Number analyzed (Participants) | 125 | 125 | 250
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 125 | 125 | 250
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 32.1 (12.6) | 31.6 (11.6) | 31.9 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67 | 67 | 134
  Male | 58 | 58 | 116
Region of Enrollment [Number; unit: participants]
  Germany | 125 | 125 | 250

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline Sore Throat Pain Intensity
Description: 100 milimeter (mm) visual acuity score (left=no pain=0mm, right=worst possible pain=100mm)
Time Frame: Baseline and 2 hours post-dose
Population: Intent to treat
Measure: Mean (95% Confidence Interval); unit: mm
Arm/Group | Lidocaine 8mg +CPC 2mg | Lidocaine 1mg + CPC 2mg
Number analyzed (Participants) | 125 | 125
mm | -27.4 [-31.0 to -23.8] | -26.9 [-30.5 to -23.3]

2. Secondary Outcome: Change From Baseline Sore Throat Pain Intensity up to 240 mn Post-dose
Description: 100 milimeter (mm) visual acuity score (left=no pain=0mm, right=worst possible pain=100mm). It measures the highest pain level felt by the patient.
Time Frame: Baseline and 240 mn post-dose
Population: intent to treat
Measure: Mean (95% Confidence Interval); unit: mm
Arm/Group | Lidocaine 8mg +CPC 2mg | Lidocaine 1mg + CPC 2mg
Number analyzed (Participants) | 125 | 125
mm | -25.5 [-29.8 to -21.2] | -29.1 [-33.1 to -25.1]

ADVERSE EVENTS:
Time Frame: 14 Dec 2010 to 5 Apr 2011
Arm/Group | Lidocaine 8mg +CPC 2mg | Lidocaine 1mg + CPC 2mg
Serious Adverse Events (participants affected / at risk) | 1/125 | 0/125
Other Adverse Events (participants affected / at risk) | 10/125 | 9/125
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lidocaine 8mg +CPC 2mg (N=125) | Lidocaine 1mg + CPC 2mg (N=125)
Tendon rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lidocaine 8mg +CPC 2mg (N=125) | Lidocaine 1mg + CPC 2mg (N=125)
Headache (Nervous system disorders) | 7 (7) | 6 (6)
Throat Irritation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
dizziness (Nervous system disorders) | 0 (0) | 1 (1)
hyperaesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Stridor (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
vertigo (Nervous system disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Preliminary agreement between Novartis Consumer Health and the investigator